CLINICAL TRIAL: NCT04168203
Title: Randomized Controlled Trial of Extended-Duration Low-Intensity Apixaban to Prevent Recurrence in High-Risk Patients With Provoked Venous Thromboembolism
Brief Title: Extended-Duration Low-Intensity Apixaban to Prevent Recurrence in High-Risk Patients With Provoked Venous Thromboembolism
Acronym: HI-PRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV185-745
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Venous Thromboembolism
Keywords: pulmonary embolism; deep vein thrombosis; venous thromboembolism; secondary prevention; anticoagulation
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: 600-patient U.S.-based, single-center, randomized, double-blinded, placebo-controlled study of apixaban 2.5 mg orally twice daily for extended prevention of recurrence after provoked VTE in patients with at least one persistent provoking factor who have completed at least 3 months of standard therapeutic anticoagulation and who have a low risk of bleeding.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Extended Duration Thromboprophylaxis (Experimental): apixaban 2.5 mg orally twice daily for a duration of 12 months
  Interventions: Drug: Apixaban 2.5 MG
- Control (Placebo Comparator): oral placebo for a duration of 12 months
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Apixaban 2.5 MG — apixaban 2.5 mg orally twice daily for a duration of 12 months
  Arms: Extended Duration Thromboprophylaxis
Drug: Placebo oral tablet — placebo oral tables twice daily for a duration of 12 months
  Arms: Control

SUMMARY:
Design: U.S.-based, single-center, randomized placebo-controlled trial.

Brief Treatment Description: Low-intensity apixaban (2.5mg twice daily) for extended-duration secondary prevention of VTE after initial treatment for provoked VTE.

Purpose: To establish the safety and efficacy of low-intensity apixaban versus placebo for extended prevention of recurrence after provoked VTE in patients with at least one persistent provoking factor.

Population: Outpatients with provoked VTE with at least one persistent provoking factor.

Enrollment: 600 subjects

Randomization: 1:1

Clinical Site Locations: 1 center (Brigham and Women's Hospital)

Study Duration: 36 months; enrollment period of up to 20 months with 12-month follow-up.

Primary Safety and Efficacy Outcomes:

Primary Safety Outcome: International Society on Thrombosis and Haemostasis (ISTH) major bleeding at 12 months.

Primary Efficacy Outcome: Symptomatic, recurrent VTE, defined as the composite of deep vein thrombosis and/or pulmonary embolism at 12 months.

Secondary Efficacy Outcome: The composite of death due to cardiovascular cause, nonfatal myocardial infarction, stroke or systemic embolism, critical limb ischemia, or coronary or peripheral ischemia requiring revascularization (major adverse cardiovascular events, including major adverse limb events) at 12 months.

Follow-Up: Follow-up will consist of Electronic Health Record (EHR) review at 12-months from study enrollment.

Interim Analysis: An interim analysis for the primary safety and efficacy outcomes will be performed when 300 subjects have completed 12-month follow-up.

DETAILED DESCRIPTION:
Provoked venous thromboembolism (VTE) is traditionally considered a transient acute disorder requiring a limited duration of anticoagulant therapy. Patients who suffer deep vein thrombosis (DVT) or pulmonary embolism (PE) following major surgery, major trauma, or periods of immobility are generally treated with time-limited anticoagulation for 3 months. However, provoked VTE patients have recently been recognized as a heterogeneous population comprised of those with transient provoking and persistent provoking risk factors (1). Common risk factors in provoked VTE such as obesity, immobility, atherosclerotic cardiovascular disease, heart failure, chronic lung disease, chronic kidney disease, and inflammatory disorders frequently contribute to an enduring rather than transient risk. Furthermore, epidemiological studies (8,9) and the randomized clinical trial EINSTEIN CHOICE (3) suggest that VTE is best characterized as a chronic disorder with periodic relapses. A landmark Danish National Registry analysis demonstrated that patients who suffer provoked or unprovoked VTE have an increased risk of recurrence over the ensuing 30 years and that recurrent PE causes increased mortality (10). While the rate of VTE recurrence ranges 30-50% over 10 years for unprovoked VTE (also termed idiopathic; unprovoked implies that an immediate trigger for the VTE cannot be identified), recurrent events occur in about 20% of patients over 10 years after a provoked event (provoked VTE is defined as post-operative, post-major trauma, post-hospitalization, or related to pregnancy, hormonal contraception/replacement therapy, or immobility) (11-13). Based on these data, provoked VTE patients represent a population vulnerable to VTE recurrence, especially at the transition of care from the initial (acute) treatment phase to the chronic treatment phase, at which point anticoagulation is discontinued in most of these patients.

The EINSTEIN CHOICE trial recently evaluated the safety and efficacy of regimens of full- or lower-intensity anticoagulant therapy versus low-dose aspirin for secondary prevention of VTE after an initial provoked or unprovoked event (2). The EINSTEIN CHOICE Investigators randomly assigned 3396 patients with VTE to receive either once-daily rivaroxaban (at doses of 20 mg or 10 mg) or 100 mg of aspirin. Prior to enrollment in EINSTEIN CHOICE, all study patients completed 6 to 12 months of anticoagulation therapy, and their providers were in equipoise regarding the need for extended anticoagulation. Approximately 60% of patients in EINSTEIN CHOICE had suffered provoked VTE. Symptomatic recurrent VTE occurred in 17 of 1107 patients (1.5%) receiving 20 mg of rivaroxaban and in 13 of 1127 patients (1.2%) receiving 10 mg of rivaroxaban, and in 50 of 1131 patients (4.4%) receiving low-dose aspirin (hazard ratio for 20 mg of rivaroxaban vs. aspirin, 0.34; 95% confidence interval [CI], 0.20 to 0.59; hazard ratio for 10 mg of rivaroxaban vs. aspirin, 0.26; 95% CI, 0.14 to 0.47; P<0.001 for both comparisons). Rates of major bleeding were similar (0.5% in the group receiving 20 mg of rivaroxaban, 0.4% in the group receiving 10 mg of rivaroxaban, and 0.3% in the low-dose aspirin group) (2).

Data from 4,553 patients in EINSTEIN CHOICE and the EINSTEIN VTE Continued Treatment Study demonstrate that provoked VTE patients with persistent provoking factors have a reduction in recurrence with extended duration anticoagulation compared with low-dose aspirin or placebo (1.5% vs. 4.9%) (2,3). Common persistent provoking factors included immobility, obesity, heart failure, and chronic inflammatory disorders, such as Crohn's Disease and rheumatoid arthritis. Despite being highly prevalent, persistent provoking factors are rarely considered when stopping anticoagulation in patients with provoked VTE who have completed the typical 3- to 6-month duration of therapy. The 2016 American College of Chest Physicians (ACCP) Guidelines on Antithrombotic Therapy for VTE do not distinguish between transient and persistent provoking risk factors and recommend limited-duration anticoagulation for provoked events (4).

However, an emerging opinion is that optimal duration of anticoagulation in provoked VTE patients should be determined based on data from the extended duration rivaroxaban trials (5). Such a strategy breaks from the tradition of dichotomizing VTE as provoked or unprovoked. Rather, persisting risk factors such as heart failure, obesity, family history of VTE, acquired or hereditary thrombophilia, and immobilization are incorporated into the decision-making process for pathways focused on secondary prevention.

A suitable long-term strategy for secondary prevention has been recommended in evidence-based clinical practice guidelines for patients with unprovoked VTE (4). Extended-duration anticoagulation with warfarin or the direct oral anticoagulants (DOACs) is validated and recommended for prevention of recurrent unprovoked VTE in patients with a low-risk of bleeding (6). However, current evidence-based clinical practice guidelines are inadequate for secondary prevention in patients with provoked VTE based on several extended-duration anticoagulation trials that included patients with provoked and unprovoked VTE. In a randomized controlled trial of rivaroxaban for extended-duration secondary prevention in patients with either provoked (26%) or unprovoked (74%) DVT, recurrent VTE occurred in 8 patients (1.3%) in the rivaroxaban group compared with 42 patients (7.1%) in the placebo group (hazard ratio, 0.18; 95% CI, 0.09 to 0.39; P<0.001, relative risk reduction, 82%) (3).

In a landmark extension trial of patients with unprovoked VTE, the AMPLIFY-EXT trial compared two doses of apixaban (2.5 mg and 5 mg, twice daily) with placebo in 2486 patients with VTE who had completed 6 to 12 months of anticoagulation therapy and for whom there was clinical equipoise regarding the need for extended-duration anticoagulant therapy for secondary prevention (7). Symptomatic recurrent VTE or death from VTE occurred in 73 of the 829 patients (8.8%) who were receiving placebo versus 14 of the 840 patients (1.7%) who were receiving 2.5 mg of apixaban and 14 of the 813 patients (1.7%) who were receiving 5 mg of apixaban (p<0.001 for both comparisons). In Kaplan-Meier analysis, the apixaban 2.5 mg twice daily regimen demonstrated a major and clinically-relevant nonmajor bleeding rate similar to that of placebo. While approximately 9% of the patients in the AMPLIFY-EXT trial had transient or reversible risk factors for VTE, the provoked VTE population only accounted for approximately 200 patients and precluded a well-powered analysis. Furthermore, the intent of the AMPLIFY-EXT trial was to study unprovoked VTE (7). Finally, the HI-PRO trial is evaluating a more complex aspect of VTE secondary prevention. Rather than using the simple dichotomized view of VTE as provoked or unprovoked, HI-PRO is focusing on how the risk of recurrence in patients with persisting provoking factors may be modulated by low-dose apixaban. The foundation of this question is based on the current direction in which the field of VTE is moving (5) and supported by the more pathophysiologically-sound ISTH classification of risk factors (1).

Apixaban 2.5 mg twice daily may have additional advantages for extended-duration secondary prevention of VTE compared with rivaroxaban 10 mg daily (which has U.S. FDA approval for extended-duration therapy). Apixaban is a more pharmacokinetically rational regimen, given the half-life of these two DOACs. In trials of stroke prevention of atrial fibrillation, apixaban demonstrated a relatively lower frequency of gastrointestinal bleeding compared with warfarin (14-17). Apixaban has fewer off-target side effects than rivaroxaban, which can cause severe headache (necessitating urgent head CT) and severe rash.

Based on the emerging evidence that provoked VTE patients may require extended-duration anticoagulation for secondary prevention, the apixaban 2.5 mg twice daily dose could be a critical addition to our armamentarium in those at high risk for recurrence at the transition of care from the acute to the chronic treatment phase. However, this hypothesis needs to be tested in a clinical trial. The proposed study is a single-center, randomized controlled trial conducted at Brigham and Women's Hospital (BWH) to evaluate the feasibility of low-intensity apixaban (2.5 mg twice daily) in a study population exclusively comprised of provoked VTE patients with persistently provoking risk factors for VTE.

The study has the following specific aims:

Specific Aim #1: To compare the 12-month rate of recurrent symptomatic VTE in patients with provoked VTE and at least one persistent provoking factor who are randomized to either apixaban (2.5 mg orally twice daily) as monotherapy or placebo after completing at least 3 months of therapeutic anticoagulation and who have a low risk of bleeding.

Hypothesis #1: Compared with placebo, oral apixaban (2.5 mg twice daily) will reduce the 12-month rate of symptomatic VTE in patients with provoked VTE and at least one persistent provoking factor who have completed at least 3 months of therapeutic anticoagulation and who have a low risk of bleeding.

Specific Aim #2: To compare the 12-month rate of ISTH major bleeding in patients with provoked VTE and at least one persistent provoking factor who are randomized to either apixaban (2.5 mg orally twice daily) as monotherapy or placebo after completing at least 3 months of therapeutic anticoagulation and who have a low risk of bleeding.

Hypothesis #2: Compared with placebo, oral apixaban (2.5 mg twice daily) will be associated with a similar rate of ISTH major bleeding at 12 months in patients with provoked VTE and at least one persistent provoking factor who are randomized to either apixaban (2.5 mg orally twice daily) as monotherapy or placebo after completing at least 3 months of therapeutic anticoagulation and who have a low risk of bleeding.

Study Design

600-patient U.S.-based, single-center, randomized, double-blinded, placebo-controlled study of apixaban 2.5 mg orally twice daily for extended prevention of recurrence after provoked VTE in patients with at least one persistent provoking factor who have completed at least 3 months of standard therapeutic anticoagulation and who have a low risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Age ≥ 18 years
* Objectively-confirmed provoked DVT and/or PE
* Treated for at least 3 months with standard therapeutic anticoagulant therapy
* Has not suffered symptomatic recurrence during prior anticoagulant therapy
* Outpatient follow-up at BWH
* AND have at least one of the following persistent provoking VTE risk factors:

  * Persistent immobility (defined as paralysis, other inability to ambulate freely, bed-bound, wheelchair-bound)
  * Obesity (defined as BMI ≥ 30 kg/m2)
  * Heart failure (systolic, diastolic, or combined)
  * Chronic lung disease (COPD, asthma, interstitial lung disease)
  * Chronic kidney disease (nephrotic/nephritic syndrome, renal dysfunction with creatinine ≤ 2.5 mg/dL)
  * Chronic inflammatory/autoimmune disorder (inflammatory arthritis, vasculitis, inflammatory bowel disease, chronic infection)
  * Atherosclerotic cardiovascular disease (coronary, cerebrovascular, or peripheral artery disease) (up to 35% in each study group may have atherosclerotic cardiovascular disease as a qualifying persistent risk factor)
  * NOTE: Eligible patients will be allowed to have multiple risk factors, and there will not be a limit as to how many of the above risk factors a subject may have. In addition, we will place no limit on the number of patients included with multiple risk factors. A study population with multiple risk factors is highly representative of the provoked VTE population and will provide the greatest generalizability of the study results to real-world clinical practice. Including patients with single and multiple persistent provoking risk factors will also facilitate enrollment. As noted, there is clinical and research equipoise regarding whether patients with a single or multiple persistent provoking VTE risk factors should receive extended duration thromboprophylaxis for secondary prevention.
* Willing to provide written informed consent

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control (such as oral contraceptives, other hormonal contraceptives [vaginal products, skin patches, or implanted or injectable products], or mechanical products such as an intrauterine device or barrier methods [diaphragm, condoms, spermicides]) to avoid pregnancy for the entire study
* Active cancer within the past 5 years
* Contraindication to antithrombotic or antiplatelet therapy
* Requirement for ongoing anticoagulant therapy, dual antiplatelet therapy, P2Y12 inhibition, or aspirin at a dose of > 81 mg daily
* Hemoglobin level < 9 mg/dL, a platelet count < 100,000/mm3, a serum creatinine level > 2.5 mg/dL, an ALT or AST level > 2 times the upper limit of the normal range, or a total bilirubin level > 1.5 times the upper limit of the normal range
* History of bleeding diathesis or have had recent active bleeding
* Active severe hepatobiliary disease
* More than 6 months that have elapsed without taking an anticoagulant or low-dose aspirin

  o NOTE: The risk of recurrent VTE following cessation of anticoagulation rises slowly over the first 3-6 months (26). After this initial period, the cumulative risk of recurrent VTE steepens. Using a limit of no greater than 6 months of interruption in anticoagulation before potential reinitiation of anticoagulation as part of this trial will safely facilitate enrollment as opposed to restricting the population to no greater than 3 months of interruption.
* Known severe thrombophilia (any increased titer antiphospholipid antibody or positive lupus anticoagulant/DRVVT or deficiency of antithrombin, protein C, or protein S) which would indicate long-term full therapeutic anticoagulation with a vitamin K antagonist
* Life expectancy < 12 months or hospice care
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
* Receiving concurrent non-FDA-approved or investigational agents or has received an investigational agent within the past 30 days prior to the first dose of study treatment (with the exception of approved medications being used for an approved indication, e.g., investigating a new dosing regimen for an approved indication)
* Any condition, which in the opinion of the investigator, would put the subject at an unacceptable risk from participating in the study
* Any other medical, social, logistical, or psychological reason, which in the opinion of the investigator, would preclude compliance with, or successful completion of, the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Derived] Piazza G, Bikdeli B, Pandey AK, Krishnathasan D, Khairani CD, Bejjani A, Morrison RH, Hogan H, Rashedi S, Pfeferman M, Lou J, Fanikos J, Porio N, Rosenbaum L, Sobieszczyk P, Lan Z, Gerhard-Herman M, Campia U, Goldhaber SZ; HI-PRO Trial Investigators. Apixaban for Extended Treatment of Provoked Venous Thromboembolism. N Engl J Med. 2025 Sep 25;393(12):1166-1176. doi: 10.1056/NEJMoa2509426. Epub 2025 Aug 30. PMID 40888734

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Duration Thromboprophylaxis | Control
Started | 300 | 300
Completed | 300 | 300
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Duration Thromboprophylaxis | Control | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 200 | 200 | 400
  >=65 years | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (15.2) | 59.9 (15.2) | 59.5 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 166 | 342
  Male | 124 | 134 | 258
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 37 | 70
  White | 246 | 239 | 485
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 16 | 20 | 36
Region of Enrollment [Number; unit: participants]
  United States | 300 | 300 | 600

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Symptomatic, Recurrent VTE Defined as the Composite of Deep Vein Thrombosis and/or Pulmonary Embolism
Description: DVT is diagnosed as a newly non-compressible venous segment or segments on ultrasonography or a filling defect on computed tomographic (CT) venography, magnetic resonance (MR) venography, or contrast venography.
  PE is diagnosed based on new mismatched perfusion defect(s) on ventilation perfusion scan, the presence of a new pulmonary artery filling defect on contrast-enhanced chest CT, a new finding of intraluminal filling defect on invasive pulmonary angiography, or evidence of PE at autopsy.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Duration Thromboprophylaxis | Control
Number analyzed (Participants) | 300 | 300
Participants | 4 | 30

2. Primary Outcome: Frequency of Major Bleeding
Description: Defined as overt bleeding that is associated with a decrease in the hemoglobin level ≥ 2 g/dL, leads to transfusion ≥ 2 units of packed red blood cells, occurs in a critical site, or contributes to death
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Duration Thromboprophylaxis | Control
Number analyzed (Participants) | 300 | 300
Participants | 1 | 0

3. Secondary Outcome: Frequency of the Composite of Death Due to Cardiovascular Cause, Nonfatal Myocardial Infarction (MI), Stroke or Systemic Embolism, Critical Limb Ischemia (CLI), or Coronary or Peripheral Ischemia Requiring Revascularization
Description: An acute MI is defined as the presence of at least 2 of 3 following conditions (29):
  * Cardiac biomarkers, with at least one of the values being elevated with at least one value above the 99th percentile upper reference limit) and with at least one of the following:
  * symptoms of myocardial ischemia
  * new (or presumably new) significant ST-segment/T-wave changes or left bundle branch block
  * development of pathological Q waves on ECG
  * new loss of viable myocardium or regional wall motion abnormality by imaging
  * identification of intracoronary thrombus by angiography or autopsy
  An acute stroke is defined as a new, focal neurologic deficit of sudden onset, lasting at least 24 hours confirmed by a neurologist and neuroimaging (7). Cardiovascular death is defined as a death for which a definite non-cardiovascular cause (e.g. cancer) has not been identified.
  Major adverse limb events include acute limb ischemia (ALI) and critical limb ischemia (CLI) (30).
Time Frame: 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Frequency of Clinically Relevant Non-major Bleeding
Description: Overt bleeding that does not meet the criteria for major bleeding but that is associated with the need for medical intervention, unscheduled contact with a physician, interruption or discontinuation of the study drug, or discomfort or impairment of activities of daily living
Time Frame: 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Adherence to the Twice-daily Regimen of Apixaban (and Placebo)
Description: Total number of doses taken divided by the total number of doses prescribed
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Definitions do not differ
Arm/Group | Extended Duration Thromboprophylaxis | Control
All-Cause Mortality (participants affected / at risk) | 1/300 | 3/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300
Other Adverse Events (participants affected / at risk) | 6/300 | 6/300
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Duration Thromboprophylaxis (N=300) | Control (N=300)
Adverse Drug Reactions (General disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04168203/Prot_SAP_000.pdf